CLINICAL TRIAL: NCT05252143
Title: Elastic Properties of the Ascending Aorta Evaluated by Imaging and Biaxial Testing
Brief Title: Evaluation of Elastic Properties of Ascending Aorta
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier La Chartreuse (Other)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, Dr, Centre Hospitalier La Chartreuse
Other Study IDs: MECATHOR
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Compliance, Magnetic Resonance Imaging, Biaxial Testing, Elastic Modulus
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to assess a correlation between local patient specific elastic modulus distribution of the ascending aorta from a biaxial tensile test and MRI measurements of the elastic properties of the aorta.

A total of 70 patients referred for ascending aorta (AA) replacement underwent a preoperative cardiac-MRI for the evaluation the elastic properties and ascending aorta tissue was collected for biaxial testing to obtain maximum elastic modulus

DETAILED DESCRIPTION:
Observational and prospective trial on medical data only. The patients are operated of planned aortic aneurysm without additional intervention.

The preoperative cardiac MRI are planned in standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patient referred for ascending aorta aneurysm requiering replacement
* elective patient

Exclusion Criteria:

* claustrophobia
* contraindication to performing cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients operated in cardiac surgery unit of Dijon hospital starting in December 2018
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
aortic compliance of ascending aorta (mm2/mmHg) | preoperative cardiac MRI performing between 1 month and 1 day before surgery
  aortic compliance is a local measurement of elastic properties which is obtained with cardiac MRI images by computer processsing

SECONDARY OUTCOMES:
maximum elastic modulus (MPa) of ascending aorta | biaxial testing performing between 1 and 6 hours after procedure
  maximum elastic modulus is a local measurement of elastic properties which is obtained by biaxial testing

CONTACTS AND LOCATIONS:
Locations (1):
- Dijon University Hospital, Dijon, France